CLINICAL TRIAL: NCT01009749
Title: Computer-Delivered Motivational Intervention to Prevent Adherence Problems Among Youth Newly Recommended for HIV Medications: Project MESA (Motivational Enhancement System for Adherence)
Brief Title: Motivational Enhancement System for Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATN 072
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: HIV
Keywords: HAART; HIV; Adherence
MeSH Terms: interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MESA (Experimental)
  Interventions: Behavioral: Motivational Enhancement System for Adherence (MESA)
- MESH (Active Comparator)
  Interventions: Behavioral: Motivational Enhancement System for Health (MESH)

INTERVENTIONS:
Behavioral: Motivational Enhancement System for Adherence (MESA) — MESA is designed to increase motivation for adherence to Highly Active Antiretroviral Therapy (HAART) among youth newly recommended to begin medications.
  Arms: MESA
Behavioral: Motivational Enhancement System for Health (MESH) — Motivational Enhancement System for Health (MESH) is an attentional control providing information on nutrition and exercise.
  Arms: MESH

SUMMARY:
This is a two-phase study, consisting of the following plan:

Phase I - This is a pre-test of the feasibility and acceptability of the beta version of a computer-delivered intervention, Motivational Enhancement System for Adherence (MESA), as well as the control intervention Motivational Enhancement System for Health (MESH) at three selected AMTUs. Following analysis of the responses in Phase I and further modification of the intervention, Phase II will be initiated.

Phase II - This is a pilot, randomized, controlled trial (RCT) testing a two-session computer-delivered intervention, MESA, designed to increase motivation for adherence to Highly Active Antiretroviral Therapy (HAART) among youth newly recommended to begin medications, as well as an attention control, MESH, matched for dose and delivery format. Phase II is open to all 15 AMTUs.

ELIGIBILITY:
Inclusion Criteria:

Phase I & II, all participants

* Engaged in care at the enrolling AMTU;
* HIV-1 infection documented by a positive result on any of the following licensed tests at any time: any HIV-1 antibody test confirmed by Western blot, HIV-1 culture, HIV-1 DNA PCR, or plasma HIV-1 RNA PCR > 1,000 copies/ml;
* Age 16 to 24 years, inclusive at the time of enrollment;
* Naïve to antiretroviral therapy; NOTE: Females who have received antiretroviral therapy for the sole purpose of preventing maternal to child transmission (MTCT) will be considered antiretroviral naïve.
* Ability to understand written and/or spoken English;
* Willingness to provide signed informed consent/assent in either English or Spanish; and
* Parental or legal guardian permission, if warranted.

Phase I MESA Participants/Phase II All Participants - Recommended by a health care provider to start HAART for treatment of HIV-1 infection within the 12 weeks prior to protocol screening.

Phase I MESH Participants

- Not recommended by a health care provider to start HAART for treatment of HIV-1 infection.

Exclusion Criteria:

Phase I & II, all participants

* Known pregnancy (pregnancy testing is not required);
* Inability to understand spoken or written English;
* Visibly distraught and/or visibly emotionally unstable (e.g., exhibiting suicidal, homicidal, manic or violent behavior);
* Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with ability to give true informed consent and to adhere to the study requirements;
* Active psychiatric condition that in the opinion of the site personnel, would interfere with the ability to give true informed consent and to adhere to the study requirements;
* Acute illness that, in the opinion of the treating clinician, would interfere with the participant's ability to adhere to the protocol requirements and/or interfere with the protocol objectives; and
* Concurrent participation or participation within the previous 4 weeks, in any behavioral intervention study or program, including, but not limited to, ATN 069 and ATN 073. Permission to co-enroll into other behavioral studies or programs must be obtained from the protocol chair or designee.

Phase II, All Participants Prior participation in the Phase I MESA intervention (Phase I MESH control participants are eligible to participate).

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility and acceptability of the Motivational Enhancement System for Adherence (MESA) among HIV-infected youth newly beginning HAART; and in an attention control condition plus standard care. | 26 months
To compare levels of motivation to adhere and adherence and reductions in HIV-1 viral loads at follow-up among youth randomized to MESA plus standard care versus those randomized to MESH plus standard care. | 26 months

SECONDARY OUTCOMES:
To compare service utilization rates among youth randomized to MESA plus standard care versus those in an attention control condition plus standard care. | 26 months
To examine self-efficacy for adherence for youth randomized to MESA plus standard care compared to those in an attention control condition plus standard care. | 26 months
To assess HAART medication knowledge among youth randomized to MESA plus standard care versus those in an attention control condition plus standard care. | 26 months
To assess levels of motivation and self-efficacy for healthy eating and exercise among youth randomized to MESH plus standard care compared to those randomized to MESA plus standard care. | 26 months
To examine the levels of nutrition and exercise knowledge among youth randomized to MESH plus standard care compared to those randomized to MESA plus standard care. | 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Naar-King, PhD, Study Chair — Adolescent Trials Network
Locations (14):
- United States (13):
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - Univ of Califormia at San Francisco, San Francisco, California
  - Children's Hosp Natinal Med Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami-Jackson Memorial Medical Center, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stoger Hospital of Cook County, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York
  - Children's Hospital at Montefiore Medical Center, The Bronx, New York
  - Children's Hopsital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- See also: ATN Website — http://www.atnonline.org